CLINICAL TRIAL: NCT00133822
Title: Placebo-Controlled Trial of Risperidone Augmentation for SSRI-Resistant Civilian PTSD
Brief Title: Civilian Post-Traumatic Stress Disorder Risperidone Clinical Trial
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Janssen, LP (Industry)
Responsible Party: Principal Investigator, Barbara O. Rothbaum, PhD, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0184-2004; RIS-EMR-4005 (Other: Other)
Record Dates: First submitted 2005-08-22; First posted 2005-08-24 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Post-Traumatic Stress Disorders
Keywords: Post-Traumatic Stress Disorder; Sertraline; Risperidone
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Sertraline; Risperidone

INTERVENTIONS:
Drug: Sertraline and Risperidone

SUMMARY:
The purpose of this study is to determine whether the administration of risperidone is effective in the treatment of selective serotonin reuptake inhibitor (SSRI)-resistant post-traumatic stress disorder (PTSD) in civilians.

DETAILED DESCRIPTION:
Individuals with PTSD often experience anxiety attacks, nightmares, or repeated unwanted memories after experiencing or witnessing life-threatening events, such as serious accidents or natural disasters, or traumatic events such as physical or sexual abuse.

Risperidone has been approved by the Food and Drug Administration for the treatment of psychotic disorders and has been found helpful for PTSD and depression, but is still considered investigational for the purposes of this study.

All qualified participants will be started on sertraline (Zoloft) for eight weeks. Patients who are still symptomatic at the end of this phase, will be invited to join the second portion of the study where they will be randomly assigned to receive risperidone or placebo (sugar pill) in addition to the sertraline. Participants will be monitored regularly for medication effects, adverse events, and PTSD symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for DSM-IV PTSD for a minimum of one month duration
* Clinician-Administered PTSD Scale (CAPS) score > or = to 50
* Able to read and complete questionnaires and interviews
* Negative urine drug screen

Exclusion Criteria:

* Pregnant or nursing
* Primary psychotic disorder; psychotic disorder; or cognitive disorder.
* Prominent suicidal or homicidal ideation
* Alcohol or substance dependence within 3 months of starting study
* Primary anxiety disorder or bipolar disorder
* Patients currently being treated with antipsychotic medication
* Patients in active psychotherapy aimed at PTSD
* Combat-related PTSD

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65
Dates: Start 2004-04; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Remission of symptoms after 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Barbara O Rothbaum, PHD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory University School of Medicine, Atlanta, Georgia
  - Duke University Medical Center South, Durham, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina

REFERENCES:
- [Derived] Rothbaum BO, Killeen TK, Davidson JR, Brady KT, Connor KM, Heekin MH. Placebo-controlled trial of risperidone augmentation for selective serotonin reuptake inhibitor-resistant civilian posttraumatic stress disorder. J Clin Psychiatry. 2008 Apr;69(4):520-5. doi: 10.4088/jcp.v69n0402. PMID 18278987